CLINICAL TRIAL: NCT05880082
Title: Clinical Application of Efficacy Prediction Model Based on Epigenomics Sequencing Technology in Neoadjuvant Immunotherapy for Esophageal Cancer
Brief Title: PPIO-004 Clinical Application of Efficacy Prediction Model Based on Epigenomics Sequencing Technology in Neoadjuvant Immunotherapy for Esophageal Cancer
Acronym: PPIO-004-EC001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, WEI GUO, chief physician, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WGUO
Record Dates: First submitted 2023-05-17; First posted 2023-05-30 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — tislelizumab; Carboplatin; Cisplatin; nedaplatin

STUDY DESIGN:
Masking Description: The study was a one-arm open study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tislelizumab, Q3W with TP regimen (Experimental): Tislelizumab 200mg, Q3W, 2-4 cycles Albumin paclitaxel 240 mg/m², adjusted according to the patient Carboplatin: AUC=5 Q3W, d1 or cisplatin: 20mg/m² iv, D1-3 Q3W or Nedaplatin: 70mg d1 Q3W
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg, Q3W, 2-4 cycles Albumin paclitaxel 240 mg/m², adjusted according to the patient Carboplatin: AUC=5 Q3W, d1 or cisplatin: 20mg/m² iv, D1-3 Q3W or Nedaplatin: 70mg d1 Q3W
  Other Names: Carboplatin; cisplatin; Nedaplatin

SUMMARY:
The goal of this observational study is to learn about in potential operable esophageal cancer patients (cT1-2N + M0 and cT3NanyM0) receiving neoadjuvant therapy. The main questions it aims to answer are: Objective response rate, Major pathological response rate. Participants will receive two to four cycles of tislelizumab plus albuminpaclitaxel and platinum-based therapy

DETAILED DESCRIPTION:
Esophageal cancer is the eighth most common cancer in the world (934,870 new cases) and the sixth most common cause of cancer death (287,270 new cases). The incidence, prevalence and histological type of esophageal cancer vary by region. About 75% of cases occur in Asia, with China accounting for the highest proportion, accounting for about 50% of the total number of cases and cancer-specific deaths. According to China's National Bureau of Statistics in 2022, there were 252,500 cases of esophageal cancer and 193,900 deaths in China in 2016, making esophageal cancer the sixth most common cancer and the fifth leading cause of cancer death in the country. The etiologies of the two most common histological subtypes (esophageal squamous cell carcinoma [ESCC] and adenocarcinoma) vary widely. In the West, heavy drinking and smoking and their synergies are major risk factors for ESCC [3]. However, in low-income countries, such as parts of Asia and sub-Saharan Africa, the major risk factors for ESCC (which typically accounts for more than 90% of all esophageal cancer cases) have not been elucidated.

For subjects with locally advanced ESCC, international treatment guidelines recommend esophagectomy followed by preoperative chemoradiotherapy.

However, in the clinical practice, many subjects with locally advanced ESCC receive neoadjuvant chemotherapy rather than neoadjuvant chemoradiotherapy, due to safety concerns regarding the use of radiotherapy in neoadjuvant therapy and difficulties in cross-clinical collaboration, and may not receive the best benefit from neoadjuvant therapy. For the preoperative treatment of locally advanced esophageal cancer, preoperative chemotherapy also has a better survival benefit than surgery alone. In the Medical Research Council OEO2 study, median survival was 16.8 months in the preoperative chemotherapy group and 13.3 months in the surgery alone group, with 2-year survival rates of 43% and 34%, respectively. Long-term follow-up confirmed that preoperative chemotherapy had a survival benefit, with 5-year survival rates of 23% in the preoperative chemotherapy group and 17.1% in the surgery alone group. And data on other immune checkpoint inhibitors suggest that neoadjuvant chemotherapy combined with immunotherapy improves clinical outcomes.

PD-1 inhibitors have demonstrated significant benefits as second-line and first-line therapy for ESCC and in combination with chemotherapy for many other solid tumors. Preclinical studies have shown that the PD-1/PD-L1 axis can be activated early in solid tumors, and the preoperative induction of immune response may have a lasting protective effect. Preoperative immunotherapy is likely to be more effective given that the tumor antigen drops sharply after surgical resection and the removal of intact blood vessels and lymph nodes that deliver the drug may affect immunotherapy efficacy. Several Phase 1/2 and 2 studies have shown a controllable safety profile and preliminary demonstration of efficacy when adding PD-1/PD-L1 inhibitors to perioperative treatment in resectable EC subjects. PD-1 inhibitors have shown significant benefits in both second-line and first-line treatment. Given the evidence of antitumor activity of immunotherapy in patients with ESCC and the continuing need to improve survival and reduce recurrence rates of resectable esophageal cancer, several studies exploring the antitumor activity of immunotherapy in the treatment of resectable disease have tentatively shown promising prospects as a neoadjuvant therapy.

tislelizumab, as an innovative PD-1 inhibitor, has shown similar benefits to other PD-1 inhibitors in a variety of tumor types. Bb-a317-205 also showed preliminary antitumor activity in ESCC subjects, with a confirmed ORR of 46.7%, DCR of 80%, and DOR of 12.8 months. The median OS was 14.31 months. In addition, three pivotal Phase 3 studies in the ESCC field are underway (studies BGB-A317-302, BGB-A317-306, BGB-A317-311, and BGB-A317-213).

Therefore, the combination of neoadjuvant chemotherapy with tislelizumab may be a potential treatment option to improve the benefit of potentially resectable locally advanced ESCC subjects.

Cancer survival rates are often low, most likely due to advanced stage of diagnosis and limited access to timely and reasonable treatment. Early and accurate detection of cancer is important for clinical diagnosis, effective toxicity monitoring, and ultimately successful treatment of cancer. In the context of the current "precision medicine" concept, disease assessment should selectively obtain and extract key biological information from clinical phenotypes, pathological characteristics and molecular information of diseases, and carry out qualitative, positioning, quantitative and periodic accurate analysis of these information, laying the foundation for disease classification, clinical decision-making and prognosis. Based on accurate analysis of patients' biological information, treatment principles, rules and guidelines based on empirical evidence, combined with patients' unique physiological, psychological, social characteristics and personal will, effective treatment methods are wisely selected and integrated to form the best treatment plan that fits patients' unique characteristics.

In the context of the current "precision medicine" concept, disease assessment should selectively obtain and extract key biological information from clinical phenotypes, pathological characteristics and molecular information of diseases, and carry out qualitative, positioning, quantitative and periodic accurate analysis of these information, laying the foundation for disease classification, clinical decision-making and prognosis. At present, several prediction models for evaluating the efficacy and prognosis of patients have been developed by using public databases at home and abroad. However, due to the small sample size, less information included in the models and lack of clinical practice, the reliability is weak.

Therefore, new biomarkers need to be developed to better select patients, and the development of strong biomarkers and improved patient selection will be key to combination immunotherapy.

Objective response rate, major pathological response rate, pathological complete response rate, overall survival, progression-free survival, disease control rate, duration of response, R0 removal rate, adverse events, and potential predictive biomarkers were evaluated in patients undergoing surgery after tirelizumab combined with chemotherapy as neoadjuvant therapy. Explore potential Cancer biomarkers in patients undergoing surgery after receiving tislelizumab combined with chemotherapy as neoadjuvant therapy

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. Pathology (histology) confirmed potentially resectable stage cT1-2N + M0 and stage cT3NanyM0 ESCC (AJCC 8th edition); 3. Received tirelizumab combined with chemotherapy before surgery; 4.ECOG score: 0 or 1; 5. R0 radical excision can be performed; 6. Measurable or evaluable lesions assessed by the investigator according to RECIST version 1.1; 7. With my consent and signed informed consent, I shall comply with the planned visit, research treatment, laboratory examination and other test procedures.

Exclusion Criteria:

1. Patients with other malignant tumors;
2. Prior treatment for ESCC, including chemotherapy, radiotherapy, or prior antibody or drug therapy against PD-1, anti-PD-L1, anti-PD-L2, or any other specific T-cell costimulation or checkpoint pathway;
3. They are not eligible to receive platinum-containing double-drug chemotherapy regimen, chemoradiotherapy or surgery;
4. Patients with a history of fistulas caused by primary tumor infiltration, patients assessed by the investigator as being at high risk of fistulas or showing signs of perforation, and severe malnutrition;
5. Poorly controlled pleural effusion, pericardial effusion or ascites requiring frequent drainage (recurrence within 2 weeks after intervention)
6. Known human immunodeficiency virus (HIV) testing history or known acquired immunodeficiency syndrome (AIDS);
7. A history of interstitial lung disease, non-infectious pneumonia or poorly controlled lung disease (including pulmonary fibrosis, acute lung disease, etc.);
8. Any positive test result for hepatitis B virus or hepatitis C virus indicating the presence of a virus, such as hepatitis B surface antigen (HBsAg, Australian antigen) positive or hepatitis C antibody (anti-HCV) positive (except HCV-RNA negative);
9. Those who have a history of drug abuse and cannot abstain or have mental disorders;
10. Known history of allogeneic organ transplantation or allohematopoietic stem cell transplantation;
11. Patients who are participating in other clinical trials or participating in other clinical trials with less than 4 weeks to end;
12. Pregnant or lactating women;
13. Patients with a BMI < 18.5mg/m2 or a weight loss greater than 10% before screening;
14. Other conditions that the researchers believe will affect the progress of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Up to approximately 6 months
  From enrollment to the end of treatment at 4 weeks
Major pathological response rate | At Surgery approximately 4weeks after last treatment
  Pathological results were obtained after surgery

SECONDARY OUTCOMES:
Pathological complete response rate | At Surgery approximately 4weeks after last treatment
  Pathological results were obtained after surgery
Overall survival | Up to 24 months
  From enrollment to death
Progression-free survival | Up to 24 months
  From enrollment to Progression

CONTACTS AND LOCATIONS:
Locations (1):
- Army Medical Center of the People's Liberation Army, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No